CLINICAL TRIAL: NCT04966871
Title: A Clinical Trial of a 3-dose, 28-Day Regimen of PfSPZ Vaccine in Healthy, Malaria-Naïve, Adult Subjects to Determine Safety, Tolerability and Efficacy Against Heterologous CHMI Conducted 14, 42 or 70 Days After Immunization
Brief Title: Safety, Tolerability and Efficacy of PfSPZ Vaccine Against Heterologous CHMI in US Malaria naïve Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USSPZV6
Record Dates: First submitted 2021-06-03; First posted 2021-07-19 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Malaria
Keywords: PfSPZ Vaccine; Malaria; Plasmodium falciparum; Controlled human malaria infection
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group A (PfSPZ Vaccine; PfSPZ Challenge 7G8) (Experimental): 14 volunteers will receive 3 doses of 9 x 10^5 PfSPZ Vaccine on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 14 by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (7G8) for CHMI
- Group B (PfSPZ Vaccine; PfSPZ Challenge 7G8) (Experimental): 14 volunteers will receive 9 x 10^5 PfSPZ Vaccine on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 42 by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (7G8) for CHMI
- Group C (PfSPZ Vaccine; PfSPZ Challenge 7G8) (Experimental): 14 volunteers will receive 9 x 10^5 PfSPZ Vaccine on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 70 by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (7G8) for CHMI
- Group A controls (Saline; PfSPZ Challenge 7G8) (Placebo Comparator): 4 volunteers will receive Normal Saline (NS) as placebo on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 14 by DVI injection.
  Interventions: Biological: PfSPZ Challenge (7G8) for CHMI; Other: Normal Saline
- Group B controls (Saline; PfSPZ Challenge 7G8) (Placebo Comparator): 4 volunteers will receive Normal Saline (NS) as placebo on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 42 by DVI injection.
  Interventions: Biological: PfSPZ Challenge (7G8) for CHMI; Other: Normal Saline
- Group C controls (Saline; PfSPZ Challenge 7G8) (Placebo Comparator): 4 volunteers will receive Normal Saline (NS) as placebo on days 1, 8, 29.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (7G8) will be administered on day 70 by DVI injection.
  Interventions: Biological: PfSPZ Challenge (7G8) for CHMI; Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Metabolically active, non-replicating, radiation attenuated, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Vaccine)
  Arms: Group A (PfSPZ Vaccine; PfSPZ Challenge 7G8); Group B (PfSPZ Vaccine; PfSPZ Challenge 7G8); Group C (PfSPZ Vaccine; PfSPZ Challenge 7G8)
Biological: PfSPZ Challenge (7G8) for CHMI — Live, infectious, aseptic, purified, vialed, cryopreserved, Plasmodium falciparum sporozoites, strain 7G8
Other: Normal Saline — normal saline placebo control
  Arms: Group A controls (Saline; PfSPZ Challenge 7G8); Group B controls (Saline; PfSPZ Challenge 7G8); Group C controls (Saline; PfSPZ Challenge 7G8)

SUMMARY:
This is a randomized, double blind, placebo-controlled, single site, trial of a condensed regimen of PfSPZ Vaccine administered on Days 1, 8 and 29 by direct venous inoculation (DVI) to assess safety, tolerability, immunogenicity and vaccine efficacy (VE) against heterologous controlled human malaria infection (CHMI) conducted at varying time intervals after the third immunization (14, 42 or 70 days). The trial is designed to simulate pre-deployment immunization of military personnel. Prior studies with this regimen show high level protection (>80%) against CHMI at 21 days, but the onset and duration of protection have not been fully defined.

DETAILED DESCRIPTION:
USSPZV6 is a single site, double-blind, randomized, placebo-controlled, clinical trial. Study groups will be randomized in a 14:4 ratio (vaccine to NS placebo) among healthy, malaria-naive adults aged 18-50 years. There will be three groups of subjects. Each of the 3 groups will have 14 subjects who receive 3 injections with 9 x 10^5 PfSPZ of PfSPZ Vaccine and 4 subjects who receive 3 injections with normal saline placebo. Subjects who complete all immunizations will receive a total 2.7 x 10^6 PfSPZ. VE will be assessed by exposure to PfSPZ Challenge (7G8) (cryopreserved infectious sporozoites originating from a Pf strain isolated in Brazil, and thus heterologous to the vaccine). The day of CHMI will vary per group with Groups A, B and C receiving PfSPZ Challenge (7G8) on days 14, 42 or 70 after Vaccination 3 (V3), respectively. Direct observation will be for 30 minutes following each dose of PfSPZ Vaccine or PfSPZ Challenge. A research/safety monitor and a Safety Monitoring Committee (SMC) will provide safety oversight. Clinical study monitoring will be the responsibility of Sanaria or Sanaria's designated and authorized representative. Screening will not precede enrollment by more than 90 days. For the second and third immunizations, allowable windows are assigned. The entire study will take approximately 8 months to complete, including 2 months of recruitment because the study will be conducted in two sequential cohorts. The period of follow-up for each immunized subject and placebo controls is through 8 weeks post-CHMI. Study participation will last between 99 and 154 days (not including screening) depending upon group assignment.

Case report forms (CRFs) will serve as the repository of source documents and other relevant data for each study subject. Only information that cannot be collected initially into the CRF (for instance, EKGs and AE medical records) will first be collected onto separate source documents before transcription into the CRF. Laboratory results will be entered from source documents directly into the database.

Solicited adverse events (AEs) will be collected for 7 days after each immunization. Unsolicited AEs will be collected from the first immunization (V1) until 28 days after the third immunization (V3) and for 28 days after CHMI. Physical exams and medical history will be assessed as indicated. Safety laboratories will be collected at screening, day of V1, 14 days after V2, 7 days after V3, day of CHMI and 28 days after CHMI. Surveillance for SAEs will occur for the duration of the study. Follow-up of AEs (including SAEs) occurs until resolution or stability.

If clinical laboratories expire (meaning they were obtained greater than 90 days prior to planned enrollment), specific safety labs will be repeated for screening purposes. Safety evaluation includes an electrocardiogram (ECG) performed at screening. Subjects with abnormal cardiovascular symptoms or findings that appear clinically significant will be excluded and if appropriate, referred to a cardiologist for further evaluation.Clinical laboratory testings will be conducted by Fred Hutchinson Cancer Research Center.

Detection of parasitemia post CHMI will be based upon qRT-PCR. Subjects who have 2 positive qRT-PCR results separated by greater than or equal to 12 hours or a single qRT-PCR result reading > 250 estimated parasites/mL will be treated with anti-malaria therapy. Anti-malarial therapy will consist of: First-line: Malarone, Second-line: Coartem.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant female) 18 to 50 years of age
* Able and willing to participate for the duration of the study
* Able and willing to provide written (not proxy) informed consent
* Physical examination and laboratory results without clinically significant findings
* Individuals of childbearing potential must agree to use effective means of birth control (e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) during the entire study. Female participants with a history of surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other) must provide written documentation of the procedure from a health care provider
* Willing to refrain from blood donation for 3 years following CHMI
* Agree not to travel to a malaria endemic region during the entire course of the trial

Exclusion Criteria:

* A history of malaria infection within 2 years prior to study participation or travel to a malaria endemic region within six months prior to first immunization
* Receipt of a malaria vaccine in a prior clinical trial
* History of a splenectomy or sickle cell disease
* History of a neurologic disorder (including non-febrile seizures or complex febrile seizures) or formal history of migraine headache
* Current use of systemic immunosuppressant pharmacotherapy
* Receipt of a live vaccine within 4 weeks of first immunization or of a non-live vaccine within 2 weeks of first immunization
* Individuals who are breast-feeding, pregnant or planning to become pregnant during the study period
* Known allergy to atovaquone-proguanil (Malarone®), artemether-lumefantrine (Coartem), or any component of the investigational products
* History of anaphylaxis or other life-threatening reaction to a vaccine
* Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment
* Evidence of increased cardiovascular disease risk; defined as >10% five-year risk by non-laboratory method (Gaziano, 2008)
* Plan to participate in another investigational vaccine/drug research during the study
* Plan for major surgery between enrollment until 28 days post-CHMI
* Use or planned use of any drug with anti-malarial activity that would preceed or coincide with malaria challenge.
* Anticipated use of medications known to cause drug reactions with atovaquone-proguanil or artemether-lumefantrine such as cimetidine, metoclopramide, antacids, and kaolin
* Positive HIV, HBV or HCV infection
* An abnormal electrocardiogram, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically significant abnormalities on the electrocardiogram as determined by the consulting cardiologist
* Any clinically significant deviation from the normal range in biochemistry or hematology tests measured at screening and not resolving.
* Any medical, psychiatric, social, behavioral or occupational condition or situation (including active alcohol or drug abuse) that, in the judgment of the PI, impairs the volunteer's ability to give informed consent, increases the risk to the subject of participation in the study, affects the ability of the subject to participate fully in the study, or might negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Vaccine efficacy (VE) of PfSPZ Vaccine against Pf malaria in adults | 7-28 days after CHMI
  VE computed as one minus the estimated risk ratio for Pf infection (parasitemia) detected by qRT-PCR beginning 7 days after CHMI and censoring subjects at 28 days in the "modified Intention to Treat" (mITT) population
Safety and tolerability of 3 doses of 9.0x10^5 PfSPZ of PfSPZ Vaccine- solicited AEs | Day of first immunization until 8 weeks post CHMI
  The differences in proportions of vaccinees compared to controls experiencing related solicited adverse events after vaccination.
Safety and tolerability of 3 doses of 9.0x10^5 PfSPZ of PfSPZ Vaccine- solicited AEs | Day of first immunization until 8 weeks post CHMI
  The differences in proportions of vaccinees compared to controls experiencing related unsolicited adverse events after vaccination.
Safety and tolerability of 3 doses of 9.0x10^5 PfSPZ of PfSPZ Vaccine- SAEs | Day of first immunization until 8 weeks post CHMI
  The differences in proportions of vaccinees compared to controls experiencing related serious adverse events (SAEs) after vaccination.
Safety and tolerability of 3 doses of 9.0x10^5 PfSPZ of PfSPZ Vaccine- Lab abnormalities | Day of first immunization until 8 weeks post CHMI
  The differences in proportions of vaccinees compared to controls experiencing related laboratory abnormalities after vaccination.

SECONDARY OUTCOMES:
Antibody responses to PfCSP post-immunization/CHMI and correlation with protection in vaccinees vs controls | 2 weeks post Vaccination 2 until 4 weeks post CHMI
  Antibody levels to PfCSP measured by ELISA comparing vaccinees to controls
Antibody responses to PfCSP post-immunization/CHMI and correlation with protection in protected vs unprotected vaccinees | 2 weeks post Vaccination 2 until 4 weeks post CHMI
  Antibody levels to PfCSP measured by ELISA comparing protected (no parasitemia occurring post CHMI) and non-protected (parasitemia occurring post CHMI) vaccinees.
VE between different groups with CHMI at 14, 42 or 70 days after Vaccination 3 | Day of first immunization until 8 weeks post CHMI
  VE computed as one minus the estimated risk ratio for Pf infection (parasitemia) detected by qRT-PCR beginning 7 days after CHMI and censoring subjects at 28 days in the mITT population

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States